CLINICAL TRIAL: NCT07310238
Title: The Effect of Repetitive Transcranial Magnetic Stimulation on Dual-task Performance in Patients With Parkinson's Disease
Brief Title: Dual-Task Improvement in Parkinson's Via rTMS
Acronym: rTMS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Gaziantep (Other)
Responsible Party: Principal Investigator, Halil Ibrahim ERGEN, Assistant professor, University of Gaziantep
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2022/345
Record Dates: First submitted 2025-12-16; First posted 2025-12-30 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Parkinson Disease (PD); Cognition Disorders; Gait Disorders, Neurologic; Dual Task
MeSH Terms: conditions — Parkinson Disease; Cognition Disorders; Gait Disorders, Neurologic

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active rTMS Group (Experimental): Participants receive repetitive transcranial magnetic stimulation (rTMS) applied to the left dorsolateral prefrontal cortex at 5 Hz, 120% of the resting motor threshold, for 10 sessions over two weeks.
  Interventions: Device: Active Repetitive Transcranial Magnetic Stimulation (rTMS)
- Sham Stimulation (Sham Comparator): Participants receive sham stimulation using the same coil positioning and session structure as the active rTMS group, but without active magnetic output. Sham sessions match the schedule and duration of the intervention arm.
  Interventions: Device: Sham Repetitive Transcranial Magnetic Stimulation

INTERVENTIONS:
Device: Active Repetitive Transcranial Magnetic Stimulation (rTMS) — Repetitive transcranial magnetic stimulation applied to the left dorsolateral prefrontal cortex using a figure-8 coil. Stimulation delivered at 5 Hz, 120% of the resting motor threshold, 600 pulses per session, for 10 sessions over two weeks.
  Arms: Active rTMS Group
Device: Sham Repetitive Transcranial Magnetic Stimulation — Sham stimulation performed using the same coil placement, session duration, and procedures as the active rTMS condition, but without magnetic output. Sessions matched in schedule and structure to the active intervention.
  Arms: Sham Stimulation

SUMMARY:
This study aimed to evaluate the effects of repetitive transcranial magnetic stimulation (rTMS) applied to the left dorsolateral prefrontal cortex on cognitive function and dual-task performance in individuals with Parkinson's disease. Participants completed ten rTMS sessions over two weeks or received sham stimulation. Cognitive status was assessed using the Montreal Cognitive Assessment, and mobility was evaluated through single-task and multiple dual-task Timed Up and Go tests. The study examined whether rTMS could enhance cognitive abilities and improve motor-cognitive performance, which are commonly impaired in Parkinson's disease and contribute to reduced functional independence. Findings indicated that rTMS led to improvements in cognition, single-task mobility, and complex dual-task performance. The intervention was well tolerated, and no adverse events related to the stimulation intensity were reported.

DETAILED DESCRIPTION:
Parkinson's disease often leads to declines in cognition, gait performance, and the ability to manage simultaneous cognitive-motor demands. These difficulties contribute to mobility limitations, fall risk, and loss of independence in older adults. This randomized controlled study investigates whether repetitive transcranial magnetic stimulation (rTMS) targeting the left dorsolateral prefrontal cortex can enhance cognitive function and improve single- and dual-task mobility performance in individuals with Parkinson's disease. Participants complete a two-week intervention consisting of active or sham stimulation. Standardized cognitive and functional mobility assessments are administered before and after the intervention to determine the extent of change associated with rTMS. The study is designed to provide preliminary evidence on whether neuromodulation of an executive-control region can support functional motor-cognitive interactions in this population.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of Parkinson's disease.
* Age 65 years or older.
* Currently receiving dopaminergic therapy.
* Ability to stand independently for at least 30 seconds.

Exclusion Criteria:

* Inability to walk for 2 minutes without a walking aid.
* Any contraindication to transcranial magnetic stimulation (e.g., metal implants in the head, history of seizures).
* Musculoskeletal injury or structural abnormality that could affect mobility assessment.
* Presence of another neurological disease.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 41 (Actual)
Dates: Start 2022-11-15 (Actual); Primary Completion 2025-11-15 (Actual); Study Completion 2025-11-15 (Actual)

PRIMARY OUTCOMES:
Change in Cognitive Function Measured by the Montreal Cognitive Assessment (MoCA) | Baseline and after 2 weeks of intervention
  The Montreal Cognitive Assessment (MoCA) is a validated screening tool assessing attention, executive function, memory, language, visuospatial abilities, and orientation. Scores range from 0 to 30, with higher scores indicating better cognitive performance. The outcome is defined as the change in total MoCA score from baseline to post-intervention.

CONTACTS AND LOCATIONS:
Locations (1):
- Gaziantep University, Gaziantep, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared because the study involves a small sample size from a single clinical center, and the available data contain identifiable health information that cannot be fully anonymized for public release. No data-sharing infrastructure or repository has been established for this project.